CLINICAL TRIAL: NCT04450862
Title: Development and Pilot Randomised Controlled Trial of a Self-management Intervention to Help Individuals With Pulmonary Hypertension Live Better With Anxiety
Brief Title: Anxiety Self-management Intervention for Pulmonary Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 034442
Record Dates: First submitted 2020-06-19; First posted 2020-06-30 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-06

CONDITIONS: Pulmonary Hypertension; Pulmonary Arterial Hypertension; Anxiety; Anxiety Disorders
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Participants randomised to the intervention arm will receive a CBT informed, self-help intervention for anxiety in PH. This will be based on the four factor model, which is a trans-diagnostic approach to help understanding and identify behaviour change methods (Padesky & Mooney, 1990).
  Interventions: Other: Cognitive Behavioural therapy self help intervention for anxiety
- Control arm (No Intervention): A waiting-list will be used as a control condition. If the self-management intervention is found to be acceptable and not associated with any risk, then participants in the control condition will receive the intervention.

INTERVENTIONS:
Other: Cognitive Behavioural therapy self help intervention for anxiety — The intervention will involve five key components:
  Psychoeducation - Increase awareness of how PH may affect emotional health, normalisation of difficulties, and discussion of how symptoms associated with anxiety may add to the burden of the disease.
  Cognitions - Identify and challenge negative automatic thoughts associated with anxiety.
  Coping skills - Educate and practice a range of behavioural coping methods to help participants better manage their physical symptoms associated with anxiety in PH.
  Exposure - Replace avoidance of anxiety provoking situations and activities using graded exposure.
  Relapse prevention - Focus on relapse prevention with implementation intentions and promotion of problem solving.
  Arms: Intervention arm

SUMMARY:
Pulmonary hypertension (PH) is a disorder of high blood pressure that impacts the heart and lungs. Approximately, 50% of individuals with PH experience anxiety or panic disorders. There is limited evidence on psychological treatments for anxiety in PH; however, results support the use of Cognitive Behavioural Therapy (CBT). Despite the prevalence and impact of anxiety in PH; there are no widely available and/or disease specific pathways, thus highlighting an unmet need in this population. This project aims to develop and pilot, using randomised control trial methodology, a self-management intervention for individuals with PH based on principles of CBT.

DETAILED DESCRIPTION:
Project Objectives The primary aim of this study is to develop a self-management intervention in collaboration with patient, public involvement, which will consist of experts by experience and experts by education. The intervention is aimed at helping individuals with PH to manage symptoms of anxiety.

A secondary aim of the project is to conduct a pilot randomised controlled trial investigating the aforementioned self-management intervention. More specifically, the project will explore acceptability and feasibility of the intervention itself and research methodology proposed to test its effectiveness. Qualitative and quantitative data will be collected for this purpose which will focus on: attrition rates; adherence to the intervention; participant's acceptability of the intervention and research methodology (i.e. eligibility, randomisation, emotional response, perceptions); outcome measures; recruitment and data collection procedures; and any adverse effects. Moreover, this project will investigate the preliminary efficacy of the intervention on a series of primary (anxiety symptoms - Generalised Anxiety Disorder -7) and secondary measures (depression - PHQ9); HRQoL- emphasis10); dyspnoea - dyspnoea12; perception of coping - self-mastery questionnaire; and cognitive and behavioural processes (Cognitive Behavioural Processes Questionnaire (CBPQ), so that effect sizes can be calculated and used to inform sample sizes of any future definitive trials.

Design The study will be a pilot randomised superiority trial. Participants will be randomised on a 1:1 basis to either one of two groups, (1) CBT informed self-management intervention to help manage anxiety in PH or a (2) controlled waiting-list condition. A control condition is required to control for any therapeutic gains associated with being involved in a trial. Participants will be asked to complete a series of measures pre-, post- and one month following completion of the intervention. As such, a 2 (cognitive-behavioural informed intervention or control waiting list) x 3 (pre-, post- and intervention) research design will be used. Participants or researchers will not be blinded to condition allocation (i.e. participants will be aware they may be randomised to a waiting list condition, and researchers may be contacting participants during the intervention for feedback on adherence and acceptability).

Procedure From the study advert promoted by the Pulmonary Hypertension Association, participants will be directed to a dedicated webpage for the proposed project.

From there, participants will be able to read the participant information sheet. Participants interested in talking part will be asked to click on a link that will take them to a series of questionnaire hosted by Qualtrics. Participants will first be asked to complete an eligibility form. Based on their responses, if participants are not eligible they will be informed immediately that they are unable to participate in the study. If participants are eligible, they will be asked to complete a consent form and a series of questionnaires (see below). All data entered on this page will be recorded, as it will help to inform feasibility of the inclusion/exclusion criteria (i.e. is the study excluding a large percentage of people based on a certain factor).

Participants will also be informed on the advert promoted by the Pulmonary Hypertension Association, that they can contact the lead researcher (Gregg Rawlings) to ask any additional questions about the project prior to completing the eligibility form, consent form and/or questionnaires.

Eligible participants will be randomised, using an online randomiser, to either of the two arms. The programme used to randomise will be Random.org. Those randomised to the wait-list condition will be informed that they will be contacted again in four weeks asking them to complete a series of questionnaires and again in an additional month (see below). Those in the intervention condition will be sent the CBT intervention.

Participants in the intervention condition will be instructed to work systematically through the intervention. Two weeks after the intervention is sent to participants, participants will be contacted by the lead researcher (Gregg Rawlings) to check on adherence and acceptability of the intervention using a mixed-methods structured questionnaire. Participants will be attempted to be contacted a maximum of three times. Participants will have provided prior consent to be contacted.

Four weeks following the intervention being received and one month thereafter participants will be contacted asking them to complete the outcome measures (see below). During this time, participants will be contacted asking them to complete a quantitative and qualitative questionnaire on their views of participating in the intervention. This will be hosted by Qualitrics. Participants will have provided consent to be contacted for this purpose.

Data analysis

Quantitative data:

* Descriptive statistics, and a series of independent T-tests for continuous data and chi square tests for categorical data will be used to compare participants in the two intervention arms at baseline. This will help to indicate whether randomisation was effective and inform additional analyses i.e. certain variables may need to be controlled for using ANCOVAs or ANCOVA.
* A series of independent T-tests for continuous data and chi square tests for categorical data will be used to compare participants who have dropped out versus those who completed the study. This will help to further understand acceptability and reasons for attrition.
* Descriptive statistics will be reported for rates of attrition and data collected from the feedback questionnaires.
* To explore the potential effectiveness of the intervention, a mixed ANOVA or ANCOVA analysis will be conducted with assessment (pre-, post-intervention and one-month follow) being the within subjects factors and intervention arm (self-help intervention or waitlist) being the between subject factor. This will be conducted for the primary measure and each of the secondary measures. As this is a pilot study and not testing effectiveness specifically, intent to treat analysis and Bonferroni corrections will not be performed. Cohen's d will be used to interpret observed effect sizes using the parameters discussed above. A significance level of alpha (0.05) will be adopted for all statistical analysis reported. SPSS25 will be used for all statistical analysis.
* To calculate the post-hoc power analysis to inform sample sizes of future definitive randomised controlled trials, G*Power software will be used utilising the same parameters as above (i.e. two-tailed, alpha level and 80% power) - given the assumptions of the ANOVA or ANCOVA were met and therefore the effect size is valid. This will be conducted using the results from the primary outcome measure (GAD-7) and an average size of secondary measures.

Qualitative data: Qualitative data gathered from the feedback questionnaires will be analysed using a descriptive version of thematic analysis. This will adhere to the stages outline by Braun and Clarke:

1. Become familiar with the transcripts through repeated readings - participant's responses will already be in electronic format as it is collected via Qualtrics and so transcriptions will not be needed.
2. Undertake iterative coding of each transcript re-coding each narrative as new codes emerge.
3. Collate and contrast codes to create main- and sub-themes.
4. Review the themes and discuss the findings with members of the research team.
5. Final refinement of themes identifying clear titles and selecting appropriate quotations in support of each theme.
6. Write up the report making the outcome of the analysis coherent.

ELIGIBILITY:
Inclusion Criteria:

* • Aged 18 years or over

  * Diagnosis of pulmonary hypertension - participants will be asked to self-report this information
  * Able to complete the self-report questionnaires without help from others
  * Able to give informed consent - given that participants need to be proactive in entering the study, this will be assumed.
  * Literate in English

Exclusion Criteria:

* • Significant risk issues (participants will be asked to self-report this information), for example, experiencing current thoughts of self-harm or suicide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in Generalised Anxiety Disorder-7 (GAD-7) | pre intervention, post intervention (4 weeks after) and 1 month follow up
  The Generalised Anxiety Disorder-7 (GAD-7) is a seven-item scale, self-administered screening tool and anxiety severity measure for anxiety disorders including, generalised anxiety disorder, social anxiety and panic disorder. Scores range from 0-21. A score of 0-4 indicates "no difficulties", 5-9 "mild", 10-14 "moderate" and 15-21 "severe" levels. A higher score suggests greater anxiety.

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ9) | pre intervention, post intervention (4 weeks after) and 1 month follow up
  The Patient Health Questionnaire-9 (PHQ9) is a nine-item, self-administered tool to examine severity of depression. Scores range from 0-27. A score of 0-4 indicates "no difficulties", 5-9 "mild", 10-14 "moderate", 15-19 "moderately severe" and 20 or higher "severe depression". A higher score suggests greater depression.
Change in emPHasis-10 | pre intervention, post intervention (4 weeks after) and 1 month follow up
  This is a disease-specific, health-related quality of life measure asking respondents to rate ten difficulties commonly associated with PH. Scores can range form 0-50, with a higher score indicating lower quality of life.
Change in Dyspnoea 12 (D12) | pre intervention, post intervention (4 weeks after) and 1 month follow up
  The Dyspnoea 12 (D12) will be used to examine participant's breathlessness severity. Total scores range from 0-36 with a higher score indicating worse functioning
Change in Mastery Scale | pre intervention, post intervention (4 weeks after) and 1 month follow up
  The Mastery Scale will be used to investigate participant's perception of their own ability of coping. Total scores range from 7-49 with a higher score suggesting the individual perceives himself or herself as having a greater capacity to cope
Change in Cognitive Behavioural Processes Questionnaire (CBPQ) | pre intervention, post intervention (4 weeks after) and 1 month follow up
  The Cognitive Behavioural Processes Questionnaire (CBPQ) will be used to examine participant's responses to negative cognitions, emotions and behaviours that may themselves underlie anxiety disorders. Scores range from 0-120, with higher scores suggesting lower engagement in cognitive and behavioural processes.

CONTACTS AND LOCATIONS:
Overall Officials: Gregg H Rawlings, PhD, Principal Investigator — University of Sheffield
Locations (2):
- United Kingdom (2):
  - Clinical Psychology Unit, Sheffield, South Yorkshire
  - Clinical Psychology Unit, Sheffield

IPD SHARING:
Plan to Share IPD: No
Participant's data will not be shared with researchers outside of the research team. Participants will be anonymised in all publications.

REFERENCES:
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Yorke J, Corris P, Gaine S, Gibbs JS, Kiely DG, Harries C, Pollock V, Armstrong I. emPHasis-10: development of a health-related quality of life measure in pulmonary hypertension. Eur Respir J. 2014 Apr;43(4):1106-13. doi: 10.1183/09031936.00127113. Epub 2013 Nov 14. PMID 24232702
- [Background] Yorke J, Moosavi SH, Shuldham C, Jones PW. Quantification of dyspnoea using descriptors: development and initial testing of the Dyspnoea-12. Thorax. 2010 Jan;65(1):21-6. doi: 10.1136/thx.2009.118521. Epub 2009 Dec 8. PMID 19996336